CLINICAL TRIAL: NCT02286661
Title: Outcome Assessment in the Treatment of Type A2 Fractures of the Distal Radius by Short Arm Cast Versus Long Arm Cast
Brief Title: Short-Arm Casting Effective in Type A2 Fractures in the Distal Radius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Reza Kachooei, Assistant Professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1631
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short Arm Cast (Active Comparator): Short arm cast below the elbow
  Interventions: Procedure: Casting (short arm)
- Long Arm Cast (Active Comparator): Long arm cast above the elbow
  Interventions: Procedure: Casting (long arm)

INTERVENTIONS:
Procedure: Casting (long arm) — Casting using plaster of paris after closed reduction of distal radius fracture
  Arms: Long Arm Cast
Procedure: Casting (short arm)
  Arms: Short Arm Cast

SUMMARY:
Distal radius fracture (DRF) is among the most common fractures of the long bones, which comprise one sixth of all fractures. Due to its high prevalence, effect on patients' everyday life, and cost on national health resources, its proper management is very important. The investigators performed this prospective randomized clinical trial on 100 patients with DRFs. 50 patients were treated in each group either by short or long arm cast. Patients were visited during the 6th and 18th weeks after the reduction regarding loss of reduction and possible complications.

DETAILED DESCRIPTION:
After obtaining institutional review board (IRB) approval, the investigators performed this prospective randomized clinical trial on patients with DRFs admitted in three medical centers from September 2010 to February 2011. Patients signed the consent form prior to enrolment. the investigators included the patients older than 20 years with closed distal radial physis and initial radiographic evidence of extra articular DRF with at least one non-comminuted cortex. All fractures were type A2 according to the AO classification. The investigators considered fractures with dorsal angulations of more than 20 degrees, radial shortening of more than 10 millimeters and extensive cortical comminution as unstable fractures. Patients with unstable fractures were excluded from this study. Other exclusion criteria were the existence of multiple fractures or open fracture in the affected limb or other limbs, cerebral palsy, paresthesia of the affected limb due to the pervious cerebro-vascular accidents, previous severe deformity of the affected limb, diabetes and severe osteoporosis. Th investigators also excluded patients who had less than two consecutive follow-up visits. All eligible patients signed the informed consent. One hundred four patients were eligible to be included in this study; The investigators excluded four patients, as they did not tend to participate in the process of follow-up. The investigators divided 100 remaining patients into reduction with SAC or reduction with LAC groups based on the table of random numbers.

The investigators performed plain anterior posterior (AP) and lateral radiograph of the affected wrist in all patients initially to determine fracture severity. Based on the radial height, radial inclination and palmar tilt in initial radiograph, patients were divided into two groups. There were no significant differences between the groups regarding the pre-operative fracture characteristics. Most of the fractures were reduced under local anesthesia but general anesthesia or regional block were performed for selected patients. The technique of reduction was by slight traction and counter-traction and manipulation methods. In SAC group, the investigators positioned the forearm in neutral rotation and volar-ulnar deviation. The investigators applied The cast from the metacarpophalangeal joints dorsally and proximal palmar crease volarly, extending to one inch distal to antecubital fossa anteriorly and the olecranon posteriorly. Three points and inter osseous molding was performed. The investigators did the same technique in the LAC group. Additionally, The investigators positioned the elbow in 90 degrees of flexion and extended the plaster to the middle of the arm.

The investigators performed lateral and AP radiographs of the forearm after reduction and casting and measured the radiographic parameters (radial height, radial inclination and dorsal angulations). In all cases, anatomical reduction was considered a successful reduction. Immediately after reduction, patients started active motion of the fingers and tried to elevate the limb to the level at or above the heart. The investigators examined all patients regarding compartment syndrome. Besides, they informed the patients about compartment symptoms too. Many patients were treated in an ambulatory setting and discharged after six hours observation, but some patients were hospitalized and then discharged within two days after reduction. The investigators checked the alignment radiographically during the second week after the reduction. In the suspicious cases for the loss of reduction, comparison was done with contra-lateral wrist radiography. The investigators performed repeated reduction for those cases with unacceptable displacement. The reduction was unacceptable if there was more than five millimeters of displacement or more than five degrees of angulations. The surgeons converted LAC to SAC during the fourth week and removed casts after six weeks. The patients started active and passive motion of the wrist, elbow and fingers as the cast was removed. Patients referred to the clinic during the 6th and 18th weeks after the reduction. AP and lateral plain radiography of the wrist were performed in each visit. The investigators evaluated the patients regarding loss of reduction, malunion, nonunion, carpal tunnel syndrome, compartment syndrome, limitation in elbow and forearm range of motion (ROM), number of wounds and blisters, patient's satisfaction and stability of the distal radioulnar joint. In cases with unstable distal radioulnar joint during the 6th week visit, casting was continued for three more weeks in forearm supination position. In these cases forearm ROM was examined during the 9th and 18th weeks. The investigators considered the instability of distal radioulnar joint (DRUJ) when there was tenderness on DRUJ and pain on its mobility. For assessing the forearm pronation and supination, the patient tried to range the forearm by holding a pen in the fist with the elbow at 90 degrees flexed and adducted. Limits of ROM were abnormal if there was more than 10 degrees of difference comparing with the unaffected side.

The investigators scored patients' satisfaction by using the Visual Analog Scale (VAS) at 18th week follow-up. VAS consists of ten-point from zero (extremely dissatisfied) to 10 (extremely satisfied). The independent-Samples t-test and chi square test were used for statistical analysis when appropriate. The level of significance was set at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years
* Type A2 according to the AO classification
* Closed distal radial physis
* Initial radiographic evidence of extra articular DRF
* With at least one non-comminuted cortex

Exclusion Criteria:

* Fractures with dorsal angulations of more than 20 degrees
* Radial shortening of more than 10 millimeters
* Extensive cortical comminution as unstable fractures
* Patients with unstable fractures
* Existence of multiple fractures or open fracture in the affected limb or other limbs
* Cerebral palsy
* Paresthesia of the affected limb due to the pervious cerebro-vascular accidents
* Previous severe deformity of the affected limb diabetes
* Severe osteoporosis
* Less than two consecutive follow-up visits

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 18 weeks after closed reduction
  Elbow flexion-extension and forearm supination-pronation

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 18 weeks after closed reduction and casting
  Distal radioulnar joint instability